CLINICAL TRIAL: NCT06738199
Title: Glycoprotein Matrix-Bound Iron Improves Absorption Compared to Ferrous Bisglycinate Chelate and Ferrous Fumarate: a Randomized Crossover Trial
Brief Title: Glycoprotein Matrix-Bound Iron Improves Iron Absorption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mary Hardin-Baylor (Other)
Collaborators: Pharmachem Innovations (Unknown)
Responsible Party: Principal Investigator, Lemuel W. Taylor IV, Professor, University of Mary Hardin-Baylor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: GPMiron
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Evaluation of Bioavailability of Supplemental Forms of Iron
Keywords: Bioavailability; iron; absorption; postbiotic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: lab staff that did the analysis and lead author that performed statistical analyses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- glycoprotein matrix iron (Experimental): Acute glycoprotein matrix iron was ingested to assess blood appearance levels from pre and at 30-, 60-, 90-, 120-, 180-, 240-, 300-, 360-, 420-, and 480-minutes post-ingestion.
  Interventions: Dietary Supplement: dietary iron supplementation
- ferrous bisglycinate chelate iron (Experimental): Acute ferrous bisglycinate chelate iron was ingested to assess blood appearance levels from pre and at 30-, 60-, 90-, 120-, 180-, 240-, 300-, 360-, 420-, and 480-minutes post-ingestion.
  Interventions: Dietary Supplement: dietary iron supplementation
- ferrous fumarate iron (Experimental): Acute ferrous fumarate iron was ingested to assess blood appearance levels from pre and at 30-, 60-, 90-, 120-, 180-, 240-, 300-, 360-, 420-, and 480-minutes post-ingestion.
  Interventions: Dietary Supplement: dietary iron supplementation

INTERVENTIONS:
Dietary Supplement: dietary iron supplementation — This study aimed to compare the absorption kinetics of iron bound to a glycoprotein matrix (GPM) with those of ferrous bisglycinate chelate (FBC) and ferrous fumarate (FF).

SUMMARY:
A double-blind, randomized crossover study was conducted that evaluated absorption kinetics of 3 forms of dietary supplement iron by measuring iron levels in the blood after acute ingestion.

DETAILED DESCRIPTION:
Background: The biotransformation of minerals through glycosylation by microorganisms, such as yeast or probiotics, can produce nutrients bound to a food matrix, potentially enhancing their bioavailability. This study aimed to compare the absorption kinetics of iron bound to a glycoprotein matrix (GPM) with those of ferrous bisglycinate chelate (FBC) and ferrous fumarate (FF). Methods: In a double-blind, crossover design, 17 participants ingested 11 mg of iron in one of three forms: GPM (Pharmachem Innovation, Kearny, NJ, USA), FBC (Ferrochel®, Balchem Corp., Montvale, NJ, USA), or FF (FerroPharma Chemicals Ltd, Hungary). Blood samples were collected at baseline and at 30-, 60-, 90-, 120-, 180-, 240-, 300-, 360-, 420-, and 480-minutes post-ingestion. Water intake was standardized throughout the protocol, and an iron-free snack was provided at 4 hours post-ingestion. Pharmacokinetic analysis was performed, with key outcome variables including the area under the concentration vs. time curve (iAUC), maximum concentration (Cmax), and time to maximum concentration (Tmax). The a priori significance level was set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Participants had to have a normal body weight [body mass index (BMI) of 19-24.99 kg/m2] and engage in recreational physical activity, as defined by the American College of Sports Medicine guidelines.
* Participants must be healthy and have no diagnosed chronic disease conditions

Exclusion Criteria:

* Participants were not allowed to consume any nutritional supplements known to affect the measures of the current study for at least 6 weeks prior to participation, including pro-, post- and prebiotics, as well as digestive enzymes.
* Individuals who were currently being treated for or diagnosed with a gastrointestinal, cardiac, respiratory, circulatory, musculoskeletal, metabolic, immune, autoimmune, psychiatric, hematological, neurological, or endocrinological disorder.
* Participants whose body mass had deviated by more than 2% in the previous 30 days
* Participants who were unwilling to abstain from alcohol, nicotine, and caffeine for 12 hours prior to each visit.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-04-22 (Actual); Study Completion 2024-04-22 (Actual)

PRIMARY OUTCOMES:
plasma iron levels | 8 hour absorption period.
  Blood levels were assessed to determine if absorption rates were different between the 3 arms (forms of iron). Blood samples were taken at 30-, 60-, 90-, 120-, 180-, 240-, 300-, 360-, 420-, and 480-minutes post-ingestion.

CONTACTS AND LOCATIONS:
Locations (1):
- Human Performance Lab, Belton, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual data is available upon reasonable request based on the data in the actual peer-reviewed paper
Supporting Information: Study Protocol, SAP
Time Frame: From date of possible manuscript publication and 2 years following that publication date.
Access Criteria: Research can contact the listed corresponding author in published manuscript of this data.